CLINICAL TRIAL: NCT05677334
Title: Study on the Efficacy and Safety of Henagliflozin Combined with Continuous Subcutaneous Insulin Infusion in the Treatment of Type 2 Diabetes Mellitus Based on Continuous Glucose Monitoring System
Brief Title: Combination of Henagliflozin and Continuous Subcutaneous Insulin Infusion in T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K148-01
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Type2diabetes
Keywords: Continuous subcutaneous insulin infusion; sglt2i; Continuous Glucose Monitoring; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Henagliflozin+ Continuous Subcutaneous Insulin Infusion (Experimental): Combination therapy of Henagliflozin and Continuous Subcutaneous Insulin Infusion
  Interventions: Drug: Henagliflozin; Device: Continuous Subcutaneous Insulin Infusion
- Continuous Subcutaneous Insulin Infusion (Active Comparator): Continuous Subcutaneous Insulin Infusion therapy alone
  Interventions: Device: Continuous Subcutaneous Insulin Infusion

INTERVENTIONS:
Drug: Henagliflozin — Combination therapy of Henagliflozin and Continuous Subcutaneous Insulin Infusion
  Other Names: Continuous Subcutaneous Insulin Infusion
  Arms: Henagliflozin+ Continuous Subcutaneous Insulin Infusion
Device: Continuous Subcutaneous Insulin Infusion — Continuous Subcutaneous Insulin Infusion therapy alone

SUMMARY:
The Multi-center, randomized, controlled clinical trial investigate the efficacy and safety of Henagliflozin combined with continuous subcutaneous insulin infusion in newly diagnosed type 2 diabetes

DETAILED DESCRIPTION:
The therapeutic mechanisms of Sglt2i and continuous subcutaneous insulin infusion (CSII) are complementary. We hypothesized that for newly diagnosed type 2 diabetes (T2DM) with severe hyperglycemia, combination treatment with Henagliflozin and CSII could achieve glycaemic control in a shorter time, shorten the duration of hospitalization and reduce the total insulin dosage. We also hope to investigate the safety of sglt2i in combination with CSII in T2DM based on continuous glucose monitoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as type 2 diabetes mellitus, diagnosis time ≤ 2 years
2. Age between 20 and 70 years
3. Continuous use of any hypoglycemic drug ≤ 7 days within 6 months
4. 9% ≤ HbA1c ≤ 14% or fasting blood glucose ≥ 11.1 mmol/L
5. Body mass index (BMI) of between 20 and 32 kg/m2
6. Be able to understand the contents and methods of this study and sign the informed consent form voluntarily

Exclusion Criteria:

1. Diabetic ketosis or ketoacidosis, diabetic hypertonic state, diabetic lactic acidosis and other acute diabetic complications or serious chronic diabetic complications
2. Urinary tract infection or/and genital infection with clinical significance, or repeated urinary tract infection or/and genital infection history
3. Serious trauma or acute infection occurred within 4 weeks that may affect blood glucose control
4. People with negligent compensatory heart failure (NYHA grade III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, serious arrhythmia, cardiac surgery or vascular reconstruction within 6 months
5. Serious blood system disease (such as aplastic anemia, myelodysplastic syndrome) or any disease causing hemolysis or erythrocyte instability (such as malaria, hemolytic anemia)
6. Severe chronic gastrointestinal diseases, or those who have received treatment that may affect drug absorption (such as gastrointestinal surgery)
7. Uncontrolled hyperthyroidism
8. Those who have mental or nervous system diseases and are unwilling to communicate or cannot fully understand and cooperate
9. Pregnant or lactating women
10. ALT>3.0x ULN and/or AST>3.0x ULN and/or Tbil>2.0x ULN Blood ketone body>ULN eGFR<30ml/min/1.73 m2 Blood creatine kinase>3.0x ULN

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Time percentage (% TIR) in the range of 3.9~10.0 mmol/L blood glucose | Monitoring 5-14 days
  Compare the TIR of the two treatment groups

SECONDARY OUTCOMES:
Time taken for TIR >70% | 5-14 days after treatment
  Compare the time required for TIR >70% of the two groups
Mean Amplitude of Glycemic Excursions (MAGE) | 5-14 days after treatment
  Compare the mage of the two treatment groups
time below range (TBR) | 5-14 days after treatment
  Compare the TBR of the two treatment groups
total insulin dosage | 5-14 days after treatment
  Compare the total insulin dosage of the two treatment groups
time above range (TAR) | 5-14 days after treatment
  Compare the TAR of the two treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables.figures, and appendices) will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  Investigators could contact the corresponding author. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Wu Y, Huang Z, Qin Y. Efficacy and safety of henagliflozin combined with continuous subcutaneous insulin infusion in the treatment of Chinese inpatients with type 2 diabetes mellitus based on a continuous glucose monitoring system: protocol of a multicentre, open-label, inpatient, randomised, controlled trial. BMJ Open. 2024 Oct 11;14(10):e084834. doi: 10.1136/bmjopen-2024-084834. PMID 39395826